CLINICAL TRIAL: NCT02913417
Title: A Feasibility Study of Sequential Hepatic Internal Radiation and Systemic Ipilimumab and Nivolumab in Patients With Uveal Melanoma Metastatic to Liver.
Brief Title: Yttrium90, Ipilimumab, & Nivolumab for Uveal Melanoma With Liver Metastases
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: David Minor, MD (Other)
Collaborators: California Pacific Medical Center (Other); Jefferson Medical College of Thomas Jefferson University (Other); University of Chicago (Other)
Responsible Party: Sponsor-Investigator, David Minor, MD, Associate Director Melanoma Center, California Pacific Medical Center Research Institute
Organization: California Pacific Medical Center Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uveal Melanoma IIP
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Uveal Melanoma; Hepatic Metastases
Keywords: uveal melanoma; liver metastases
MeSH Terms: conditions — Uveal Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hepatic radiation followed by immunotherapy (Experimental): SIR-Spheres Yttrium 90 will be given by injection into the hepatic artery in two treatments, one for each lobe. 3-5 weeks later patients receive concurrent ipilimumab 1mg/kg q 3 wk x 4 and nivolumab 3mg/kg q 3 weeks x 4, all followed by nivolumab 240mg/kg q 2 weeks or 480 mg q 4 weeks until progression or 3 years
  Interventions: Device: SIR-Spheres® Yttrium 90; Drug: ipilimumab; Drug: nivolumab

INTERVENTIONS:
Device: SIR-Spheres® Yttrium 90 — Patient treatment will consist of three parts: first, selective internal radiation with SIR-Spheres Yttrium-90 microspheres with dosage per package insert , reduced to give 35cGymax to normal liver; second, concurrent ipilimumab 1mg/kg and nivolumab 1mg/kg every 3 weeks for 4 doses (immunotherapy part 1); then maintenance nivolumab at 480 every 2 weeks (immunotherapy part 2) until progression or 3 years
Drug: ipilimumab — ipilimumab 1mg/kg every 3 weeks x 4
  Other Names: Yervoy
Drug: nivolumab — nivolumab 3mg/kg every 3 weeks x 4 then 480mg q 4 weeks
  Other Names: Opdivo

SUMMARY:
Reports to date show limited efficacy of immunotherapy for uveal melanoma. Recent experimental and clinical evidence suggests synergy between radiation therapy and immunotherapy. The investigators will explore this synergy with a feasibility study of 26 patients with uveal melanoma and hepatic metastases who will receive SirSpheres Yttrium-90 selective internal hepatic radiation followed by immunotherapy with the combination of ipilimumab and nivolumab.

DETAILED DESCRIPTION:
Despite rapid improvements in the treatment of cutaneous melanoma, there has been little advance in therapy for uveal melanoma with hepatic metastases, an fatal orphan disease with no established therapy. Studies by Dr. Sato and others have described some activity for selective internal radiation with Yttrium90 microspheres (SIR-Spheres).There is limited activity as single agents for both the immunotherapy drugs ipilimumab (anti-CTLA-4) and nivolumab (anti-PD-1). In cutaneous melanoma the combination of ipilimumab and nivolumab is clearly synergistic with improvement in response rates and progression-free survival over single agents; however this has yet to be established for uveal melanoma.

Recent experimental and clinical evidence suggests additional synergy between radiation therapy and immunotherapy. This synergy seems most evident when radiation is given through large fraction stereotactic treatments or brachytherapy. The investigators will explore this synergy with a feasibility study of 18 patients who will receive SirSpheres Yttrium-90 selective internal radiation given through the hepatic artery in two treatments followed by immunotherapy with the combination of ipilimumab and nivolumab. The immunotherapy will be given with the dose and schedule that has been established and FDA-approved for cutaneous melanoma. Because of the generally low toxicity of Yttrium-90 selective internal radiation therapy the investigators feel it can be given in full dosage prior to full dosage of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of metastatic uveal melanoma.
2. Patients must have measurable disease as defined by RECIST (see Section 6).
3. Patients must have liver metastasis
4. Patients must have no more than one prior systemic therapeutic regimen. This includes chemotherapy, biologic therapy, biochemotherapy, or investigational treatment. This does not include any therapies given in the adjuvant setting. No prior anti-CTLA4 therapy. Prior anti PD-1 or anti-PDL-1 antibody therapy is acceptable.
5. No concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids.
6. Patients with prior selective internal radiation are candidates are eligible as long as they are candidates for repeat procedures and they have demonstrated progressive disease.
7. Age ≥ 18 years.
8. No known infection with HIV. Due to the mechanism of action of ipilimumab, activity and side effects in an immune compromised patient are unknown.
9. No active infection with Hepatitis B.
10. No active infection with Hepatitis C.
11. ECOG performance status 0 or 1.
12. Women must not be pregnant or breast-feeding due to unknown effects of treatments on the unborn fetus. All women of childbearing potential must have a blood test within 72 hours prior to randomization to rule out pregnancy. Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. Sexually mature females who have not undergone a hysterectomy or who have not been postmenopausal naturally for at least 24 consecutive months (i.e., who have had menses at some time in the preceding 24 consecutive months) are considered to be of childbearing potential. Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g.,vasectomy) should be considered to be of childbearing potential.
13. Patients must have the following lab values obtained < 4 weeks prior to starting treatment:

    * WBC ≥2000/uL
    * ANC ≥1500/mcL
    * Platelets ≥ 100,000/mcL
    * Hemoglobin ≥ 8g/dL
    * Creatinine ≤ 3.0 xULN
    * AST and ALT < 2.5 x ULN
    * Bilirubin ≤ 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
    * Albumin ≥ 3g/dL

Exclusion Criteria

1. Patients are excluded if they have liver tumor volume > 50%
2. Patients are excluded if they have active CNS metastases. Patients with history of CNS metastases must have MRI scans that show stability of brain metastases for 8 weeks.
3. Patients are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, or stage 1 or 2 cutaneous melanoma
4. Patients are excluded if they have a history of autoimmune disease, as follows: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]). Patients with a history of Guillain-Barre Syndrome are excluded but myasthenia gravis or psoriasis is acceptable.
5. Patients are excluded for any underlying medical or psychiatric condition which, in the opinion of the investigator, will make treatment hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
6. Patients are excluded if they have a history of prior treatment with ipilimumab or CTLA-4 inhibitor.
7. Patients are excluded if they have any concurrent medical condition requiring the use of systemic steroids (the use of inhaled or topical steroids is permitted).
8. Patients are excluded if they have had prior hepatic arterial embolization therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-10-10; Primary Completion 2022-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability of sequential selective internal radiation with Yttrium90 followed by immunotherapy with ipilimumab and nivolumab. | 5 years
  Determine the safety and tolerability of sequential selective internal radiation with Y90 followed by immunotherapy with ipilimumab and nivolumab in patients with uveal melanoma metastatic to the liver. Endpoints are CTAE determined grade 3-5 toxicities.

SECONDARY OUTCOMES:
Preliminary clinical efficacy | 5 years
  co-endpoints for this measure will be RECIST response rate and PFS
immunological changes | 5 years
  Changes in peripheral blood lymphocyte counts
Correlation of tissue markers and response to immunotherapy | 5 years
  Study of archival tumor tissue for tumor mutations, PDL-1, PDL-2, others
Explore relationship of response to immunotherapy with tumor melanin | 5years
  Correlate response with tumor production of melanin assessed by tumor density on MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: David R. Minor, M.D., Study Chair — California Pacific Medical Center Research Institute
Locations (3):
- United States (3):
  - California Pacific Medical Center, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Jefferson Medical College of Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minor DR, Kim KB, Tong RT, Wu MC, Kashani-Sabet M, Orloff M, Eschelman DJ, Gonsalves CF, Adamo RD, Anne PR, Luke JJ, Char D, Sato T. A Pilot Study of Hepatic Irradiation with Yttrium-90 Microspheres Followed by Immunotherapy with Ipilimumab and Nivolumab for Metastatic Uveal Melanoma. Cancer Biother Radiopharm. 2022 Feb;37(1):11-16. doi: 10.1089/cbr.2021.0366. Epub 2022 Jan 12. PMID 35021863